CLINICAL TRIAL: NCT06679712
Title: Development of 5-Aminolevulinic Acid (5-ALA) Based Novel Tranbroncheal Photodynamic Ablation for Peripheral Lung Malignant Tumors
Brief Title: Transbroncheal Novel PDT Peripheral Lung Tumor Ablation With 5-ALA
Acronym: 5ALA-TBPDT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Clinical Research Center, Chief of Thoracic Surgical Department, Taoyuan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYGH113004
Record Dates: First submitted 2024-10-22; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer - Non Small Cell; Lung Metastases From Any Primary
Keywords: Photodynamic therapy; Peripheral lung cancer; Transbroncheal Ablation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transbronchial PDT (Experimental)
  Interventions: Procedure: Transbronchial PDT lung tumor ablation

INTERVENTIONS:
Procedure: Transbronchial PDT lung tumor ablation — Transbronchial photodynamic therapy ablation for peripheral lung cancer

SUMMARY:
Photodynamic therapy (PDT) involves the use of special light-sensitive drugs that are selectively absorbed by cancer cells. When exposed to a specific wavelength of light, these drugs are activated within the tumor cells, triggering a free radical reaction that destroys the cancer cells. Currently, PDT is used in the treatment of early-stage lung cancer in the central airways or for advanced tumors causing airway obstruction. With advancements in medical technology, electromagnetic navigation bronchoscopy (EMB) can now be employed in a hybrid operating room (Hybrid OR) under radiological guidance to direct photodynamic therapy fibers to the tumor site for light therapy.

Our research team previously proposed a novel light transmission method, using Sodium Porfimer as the photosensitizer. In the Hybrid OR, electromagnetic navigation bronchoscopy was utilized to infuse Lipiodol into the bronchial tree, enhancing the illumination range through the optical fiber effect. Energy of 630 nm at 200 J/cm (400 mW/500 seconds) delivered through a 3 cm cylindrical laser fiber was deemed safe, with no significant acute complications observed. However, due to the low light dosage, the therapeutic outcome was suboptimal, although one case demonstrated tumor necrosis with no apparent damage to the surrounding lung tissue. A second-phase pilot clinical trial aimed at improving light energy and treatment coverage through a multi-session, multi-angle light exposure model is also proved this method is feasible and safe.

In addition to Sodium Porfimer, other photosensitizers are approved for clinical use in photodynamic diagnosis and therapy. For example, 5-Aminolevulinic Acid (5-ALA) has been approved for the treatment of brain cancer surgery. Similar to Sodium Porfimer, 5-ALA is a precursor of heme, and in certain cells (such as cancer cells and reticuloendothelial tissues) where there is a deficiency of the enzyme ferrochelatase, administering large amounts of 5-ALA or Sodium Porfimer leads to the accumulation of Protoporphyrin IX (PpIX). PpIX is a photosensitizer, and when exposed to a specific wavelength of light, it generates oxygen free radicals that destroy cancer cells, thereby producing the therapeutic effect of PDT.

We propose this clinical trial to explore the use of 5-ALA as a substitute for Sodium Porfimer in the novel PDT treatment of peripheral lung tumors. Compared to Sodium Porfimer, 5-ALA has the same therapeutic mechanism but a shorter half-life. It can be taken orally 2-4 hours before treatment, requires only one day of light protection post-procedure, and is more cost-effective. 5-ALA (Gliolan) has also been approved by the FDA for photodynamic diagnosis and treatment of brain cancer, and clinical trials in other cancers have demonstrated its safety and feasibility.

This phase 0 pilot clinical study plans to recruit six patients with peripheral malignant lung tumors (tumor diameter ≤ 30 mm). 5-ALA (Gliolan) will be used as the photosensitizer, and in the hybrid operating room, electromagnetic navigation bronchoscopy will guide a catheter to the tumor site. Lipiodol (iodized poppy seed oil) will be infused to coat the tumor, enhancing the light exposure range. The first three subjects will undergo a single-session light exposure to assess the feasibility and safety of the procedure. The remaining three subjects will receive multi-session, multi-angle light exposure to further verify the safety and effectiveness of the treatment. The findings from these subjects will serve as a reference for light energy parameters for future phase I clinical trials.

DETAILED DESCRIPTION:
The primary objective of this study is to develop an innovative photodynamic therapy (PDT) approach for the treatment of peripheral lung tumors. Current treatments for lung tumors (either primary lung cancer or metastases from other malignant tumors) include surgery, chemotherapy (including targeted and immunotherapy), and radiation therapy. The choice of treatment depends on tumor size, stage, genetic profile, and the patient's physical condition to ensure the most appropriate approach.

For early-stage peripheral lung tumors, the ongoing goal in medical technology is to develop minimally invasive treatment methods that could potentially replace existing surgical techniques, even those that are minimally invasive. Emerging treatments such as computed tomography (CT)-guided percutaneous ablation, bronchoscopic-guided radiofrequency ablation (RFA), microwave ablation, and photodynamic therapy (PDT) are under active research for minimally invasive management of malignant lung tumors without the need for incisions.

PDT uses a specialized photosensitizing drug that selectively accumulates in cancer cells. When exposed to a specific wavelength of light, the drug is activated, generating free radicals that destroy the tumor cells. Currently, PDT is applied to early-stage lung cancers of the central airways or for advanced tumors causing airway obstruction. With advancements in medical technology, electromagnetic navigation bronchoscopy (EMB) in a hybrid operating room (Hybrid OR) can guide photodynamic therapy fibers directly to the tumor site for precise treatment. There are currently three clinical trials (by Concordia in the U.S., Tokyo Medical University in Japan, and National Taiwan University Hospital) investigating PDT for lung cancer.

Initial findings from these trials suggest that PDT is safe and effective but has limitations. Though the treatment fibers can be accurately guided to the tumor, the penetration depth of light is limited, reaching only 1.5 to 2 cm in diameter. As a result, multiple guided light exposures are necessary to cover the entire tumor area to achieve complete curative resection, which increases the complexity of the procedure.

Light travels in straight lines and, when encountering tissue, undergoes three effects: penetration, absorption, and reflection, which limit its tissue penetration. In 2003, Dr. Friedberg in the U.S. proposed a novel light-exposure method. He infused high-refractive-index substances such as mineral oil into the airways, allowing the light to reflect and propagate along the bronchial walls, enabling greater tissue coverage beyond straight-line transmission. However, mineral oil can cause severe lung inflammation (lipoid pneumonia) if aspirated into the airways, limiting its clinical application.

Our research team discovered that Lipiodol, a poppy seed oil mixed with iodine ions (RI: 1.47), widely used in lymphatic imaging and hepatic tumor embolization, could be a suitable substitute for mineral oil. Lipiodol has been used for many years in airway infusion for lung tumor visualization, and while there have been reports of pneumonia as a complication, patients generally recover fully with short-term conventional treatment. Studies have shown that even when infused up to 20 ml via bronchoscopy, Lipiodol does not cause severe complications, making it a promising candidate for novel PDT methods to overcome light penetration limitations.

Based on this principle, our research team proposed using electromagnetic navigation bronchoscopy to infuse Lipiodol into the bronchial segment near peripheral lung tumors. By completely enveloping the tumor in Lipiodol, light exposure therapy applied to the proximal airway would allow the light to reach the Lipiodol-infused lung tissue, including the tumor and its supplying microvasculature and lymphatic structures. This would selectively kill the tumor and potential early micro-metastases.

We conducted a series of preclinical trials using pigs as models, demonstrating that Lipiodol can be infused into the peripheral lung tumor region via bronchoscopy. Furthermore, PDT with 200 J/cm (400 mW/cm for 500 seconds) was safe in Lipiodol-containing lung tissues.

A multicenter U.S. clinical trial (ClinicalTrials.gov Identifier: NCT02916745) is investigating PDT for peripheral lung tumors. In this trial, patients receive an intravenous injection of Photofrin (2 mg/kg) 48 hours before treatment. Using EMB and endobronchial ultrasound (EBUS), the treatment fiber is inserted into the tumor for light exposure (200 J/cm, 400 mW/cm for 500 seconds). By January 2019, five patients had been enrolled with no severe complications reported, confirming the safety and feasibility of this approach. Building on this study, our team proposed a pilot clinical trial to evaluate the safety and effectiveness of our novel PDT method for peripheral lung tumors.

From October 2021 to February 2022, three clinical cases were completed, with at least one month of follow-up indicating that the treatment was safe and feasible. All patients successfully completed the treatment without acute severe complications. One patient died six weeks post-treatment due to disease progression, unrelated to treatment complications. The limited treatment effect may be due to the low light dosage used for safety reasons, as tumor reduction was not significant in the follow-up. However, pathology from one patient showed partial tumor necrosis, and the surrounding normal lung tissue exhibited only mild inflammation, indicating that the light exposure method did not cause significant damage to normal tissue and had some therapeutic effect. Further clinical trials are needed to determine the optimal light dosage.

In the NCT02916745 trial, two cases received multiple light exposures from different angles (one case with three sessions and another with four), with no significant complications. Dr. Allison reported a case where a patient unable to undergo standard treatment received two light exposures 48 hours apart, with no complications and a positive outcome. Based on our single-session trial from 2022, which showed no complications, we are currently conducting a clinical trial with the same light dosage (confirmed not to cause thermal injury or lung damage) but employing multiple light exposures from different angles. We are also testing additional light exposure 48 hours later to determine the feasibility of this approach.

Aside from Sodium Porfimer, other photosensitizers have been approved for PDT, such as 5-Aminolevulinic Acid (5-ALA), which is approved for brain cancer surgery. Like Sodium Porfimer, 5-ALA is a precursor to heme, working through the same photodynamic mechanism. When administered, 5-ALA or Sodium Porfimer accumulates Protoporphyrin IX (PpIX) in certain cells (e.g., cancer cells), and light exposure (630 nm) activates PpIX to generate oxygen free radicals, destroying the tumor tissue. 5-ALA has been approved by the U.S. FDA and Taiwan's FDA for brain cancer surgery, with clinical trials demonstrating its safety in other cancers such as bladder and esophageal cancer.

Compared to Sodium Porfimer, 5-ALA has the same therapeutic mechanism but a shorter half-life. It can be taken orally 2-4 hours before treatment, requires only one day of post-treatment light avoidance, and is more cost-effective. This has led us to propose this clinical trial to replace Sodium Porfimer with 5-ALA for our novel PDT approach to treating peripheral lung tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathological diagnosis of malignant lung tumors (including primary lung cancer and metastatic lung cancer) in advanced or terminal stages.
* Patients for whom first- or second-line standard treatments (surgery, radiation therapy, or chemotherapy/immunotherapy/targeted therapy) have failed or who are unsuitable for standard treatments.
* Tumor size of less than or equal to 3 cm, clearly visible and assessable on chest CT scans.
* Patients whose tumors are inoperable or for whom surgery is not suitable.
* Patients in good physical condition with an ECOG (Eastern Cooperative - -Oncology Group) performance status score of 0 to 2.
* Patients capable of providing informed consent and willing to undergo regular follow-up during the trial.

Exclusion Criteria:

* Diagnosis of small cell lung cancer or non-solid malignancy.
* Tumor located in the central part of the lung.
* Previous radiation therapy to the area intended for treatment.
* Abnormal blood chemistry values.
* Chemotherapy within the past 4 weeks.
* Tumor invasion into major blood vessels.
* Allergy to porphyrins, porphyrin-related metabolites, Lipiodol, or iodine-based contrast agents.
* Plans to undergo curative surgery for lung tumors within the next 90 days.
* Patients with ophthalmologic diseases who may require a slit-lamp eye examination within the next 30 days.
* Mental illness that prevents the patient from undergoing bronchoscopy.
* Pregnant or planning to become pregnant, breastfeeding, or planning to breastfeed within 6 months after the procedure.
* Photodynamic therapy within the past month.
* Severe kidney or liver disease with abnormal renal or hepatic function.
* Plans to participate in another cancer treatment clinical trial within 3 months post-procedure.
* Patients with AIDS.
* Patients deemed unsuitable for the trial by the principal investigator or safety monitoring committee due to severe illness.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Transbronchial PDT ablation for peripheral lung tumor | minutes
  The study will track the success rate of patients completing the planned treatment steps. Each subject will undergo electromagnetic navigation bronchoscopy (EMB) to guide the injection of Lipiodol and the placement of the light-exposure fiber. The study will record the number of attempts required to correctly position the fiber at the tumor site and the total treatment time for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code